CLINICAL TRIAL: NCT04082260
Title: Signatures of Immune Reprogramming in Anti-CD52 Therapy of MS: Markers for Risk Stratification and Treatment Response
Acronym: ProgramMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: ProgramMS2017
Record Dates: First submitted 2019-08-28; First posted 2019-09-09 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- De novo patients with alemtuzumab: De novo patients prior and after alemtuzumab treatment initiation
  Interventions: Drug: Alemtuzumab Injection [Lemtrada]
- Alemtuzumab treatment: Patients under alemtuzumab treatment
  Interventions: Drug: Alemtuzumab Injection [Lemtrada]
- Extended alemtuzumab treatment: Patients requiring more than two alemtuzumab infusions
  Interventions: Drug: Alemtuzumab Injection [Lemtrada]

INTERVENTIONS:
Drug: Alemtuzumab Injection [Lemtrada] — Administration of 2 courses of alemtuzumab at an interval of 1 year. Course 1: Intravenous infusion of 12 mg alemtuzumab per day on 5 consecutive days.
  Course 2: Intravenous infusion of 12 mg alemtuzumab per day on 3 consecutive days.

SUMMARY:
Alemtuzumab is a highly effective therapy in relapse remitting multiple sclerosis (RRMS). The aim of this study is to elucidate the mechanism of action of the neuroprotective potential of alemtuzumab in RRMS. Therefore, the investigators will semi-annually analyse blood samples of RRMS patients treated with alemtuzumab up to 36 months. Using in vitro/ ex vivo assays the investigators aim to detect and characterize immune cells including their functional activity. Furthermore, the study aims to combine this analysis with clinical data (MRI, EDSS: Expanded Disability Status Scale, MSFC: Multiple Sclerosis Functional Composite) to reveal the underlining mechanism of action of alemtuzumab to further improve its efficacy and safety for present and future patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to the McDonald criteria 2010 and cranial MRI scan demonstrating white matter lesions attributable to MS within 5 years before prior to signing the informed consent form (ICF)
* Age > 18 years
* Written informed consent to study participation

Exclusion Criteria:

* Medical, psychiatric, cognitive, or other conditions that, in the Investigator's opinion, compromise the patient's ability to understand the patient information, to give informed consent, or to complete the study
* Any progressive form of MS
* Any condition that serves as a contraindication for alemtuzumab treatment
* Any disability acquired from trauma or another illness that could interfere with the evaluation of disability due to MS
* Major systemic disease or other illness that would, in the opinion of the Investigator, compromise patient safety or interfere with the interpretation of study results, e.g., current peptic ulcer disease or other conditions that may predispose to hemorrhage
* Significant autoimmune disease including but not limited to immune cytopenias, rheumatoid arthritis, systemic lupus erythematosus, other connective tissue disorders, vasculitis, inflammatory bowel disease, severe psoriasis
* Inability to undergo MRI with gadolinium administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will be patients with active RRMS, which will be rectruited in multiple KKNMS (Kompetenznetz Multiple Sklerose) centres.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Absolute and relative change of cell-counts compared to baseline of T cell subsets in the peripheral blood (every 6 months) | 36 month
  • T cell subsets:
  * CD (cluster of differentiation) 4 and CD8 positive T cells: naïve T cells, T effector cells, T memory cells, regulatory T cells
  * T-helper subsets: Th1, Th2, Th17
Absolute and relative change of cell-counts compared to baseline of B-cell subsets in the peripheral blood (every 6 months) | 36 month
  • B cell subsets:
  * Recent bone marrow emigrants, mature naïve, memory B cells
  * Plasma cells
Absolute and relative change of cell-counts compared to baseline of natural killer cells in the peripheral blood (every 6 months) | 36 month
  • Natural killer cells:
  * CD56bright, CD56dim
  * Natural killer T cells
Absolute and relative change of cell-counts compared to baseline of antigen-presenting cells in the peripheral blood (every 6 months) | 36 month
  • Antigen-presenting cells:
  * Dendritic cells: CD303+ plasmacytoid, CD11c+ and CD141+ myeloid dendritic cells
  * Monocytes and macrophages
Absolute and relative change of cell-counts compared to baseline of myeloid-derived suppressor cells in the peripheral blood (every 6 months) | 36 month
  • Myeloid-derived suppressor cells
Change from baseline in levels of markers of autoimmunity (ANA, cANCA and pANCA) in the serum (every 6 months): | 36 month
  - IFT (immunoflescence-test) of ANA, cANCA and pANCA
Change from baseline in levels of markers of autoimmunity (anti-dsDNA) in the serum (every 6 months): | 36 month
  - RIA (radioimmunoassay) of anti-dsDNA
Change from baseline in levels of markers of autoimmunity (anti-TSH-Receptor) in the serum (every 6 months): | 36 month
  - Levels of anti-TSH-Receptor (U/ml)
Change from baseline in levels of markers of autoimmunity(anti-TPO) in the serum (every 6 months): | 36 month
  - Levels of anti-TPO (U/ml)
Change from baseline in levels of markers of autoimmunity (Rheumatoid factor) in the serum (every 6 months): | 36 month
  - Levels of Rheumatoid factor (U/ml)
Change from baseline in levels of markers of autoimmunity (anti-CCP) in the serum (every 6 months): | 36 month
  - Levels of anti-CCP (U/ml)
Change from baseline in levels of markers of autoimmunity (anti-GBM) in the serum (every 6 months): | 36 month
  - Levels of anti-GBM (U/ml)
Change from baseline in levels of markers of autoimmunity (antiplatelet antibodies) in the serum (every 6 months): | 36 month
  - Levels of antiplatelet antibodies (U/ml)

SECONDARY OUTCOMES:
Functional characterization of T-cells and B cells in the peripheral blood (every 6 months) | 36 month

OTHER OUTCOMES:
Clinical related data: Analysis of MRI scans | 36 month
  - Number and location of lesions in MRI scans will be count
Clinical related data: Evaluation of disease activity and manifestation (EDSS) in comparison to baseline (every 6 months) | 36 month
  • Expanded Disability Status Scale (EDSS):
  * Scoring will be performed using standard scoring test from www.neurostatus.net.
  * EDSS is an ordinal clinical rating scale which ranges from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments. EDSS steps 1.0 to 4.5 refer to people with MS who are fully ambulatory, while EDSS steps 5.0 to 9.5 are defined by the impairment to ambulation.
Clinical related data: Evaluation of disease activity and manifestation (MSFC) in comparison to baseline (every 6 months) | 36 month
  • Multiple Sclerosis Functional Composite (MSFC):
  * MSFC will be administered according to the MSFC manual of the National MS Society.
  * In brief measurements on the impact of MS in three key clinical dimensions: leg function and ambulation, arm and hand function, and cognitive function are done. Raw scores in different measurement scales are transformed into standard comparable scores (z-scores) and an overall composite score is calculated.
Clinical related data: Observation of relapse rates | 36 month
  - Number and time of relapses will be counted

CONTACTS AND LOCATIONS:
Overall Officials: Sven Meuth, Prof., Principal Investigator — Department of Neurology with Institute of Translational Neurology, University Hospital Muenster
Locations (1):
- Department of Neurology, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bierhansl L, Ruck T, Pfeuffer S, Gross CC, Wiendl H, Meuth SG. Signatures of immune reprogramming in anti-CD52 therapy of MS: markers for risk stratification and treatment response. Neurol Res Pract. 2019 Dec 13;1:40. doi: 10.1186/s42466-019-0045-x. eCollection 2019. PMID 33324905